CLINICAL TRIAL: NCT04152174
Title: Pilot Prospective Randomized Controlled Study of Safety and Efficiency of Combined Extracorporeal Blood Purification in Neurosurgical ICU in Comparison With the Continuous Renal Replacement Therapy
Brief Title: Safety and Efficiency of Combined Extracorporeal Blood Purification in Neurosurgical ICU. Prospective RCT
Acronym: NEUROCOMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Burdenko Neurosurgery Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPI-2018-06-5
Record Dates: First submitted 2019-09-21; First posted 2019-11-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Septic Shock
Keywords: blood purification; CRRT; septic shock; neurosurgery; cytokine removal
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined extracorporeal blood purification (Experimental): CRRT with CVVHDF mode plus treatment with CytSorb adsorber
  Interventions: Procedure: Combined extracorporeal blood purification
- Control (Active Comparator): CRRT with CVVHDF mode
  Interventions: Procedure: CRRT

INTERVENTIONS:
Procedure: Combined extracorporeal blood purification — Patients receive combined extracorporeal blood purification: CRRT in CVVHDF mode with AN 69 ST set (Baxter) and hemoadsorption with Cytosorbents Corp. CytoSorb adsorber.
  Arms: Combined extracorporeal blood purification
Procedure: CRRT — Patients receive CRRT in CVVHDF mode with AN 69 ST set (Baxter)
  Arms: Control

SUMMARY:
To assess the efficiency and safety of combined extracorporeal blood purification in patients with septic shock in Neurosurgical ICU in comparison with the efficiency and safety of the continuous renal replacement therapy (CRRT).

DETAILED DESCRIPTION:
According to studies and modern sepsis treatment guidelines, conventional CRRT has not proved effective in the septic shock treatment.

Effectiveness of other extracoporeal blood purification methods, such as hemoadsorption or combined blood purification (hemoadsorption combined with CRRT) is widely pointed out in current publications: contemporary studies in general ICU patients demonstrated that the use of hemoadsorption or combined extracorporeal blood purification methods is effective for septic shock patients treatment.

It has been proven that cytokines discharged into the systemic blood flow are the key pathophysiological mechanism of septic shock. Hemoadsorption allows for significantly more effective removal of different inflammatory mediators than the traditional methods of CRRT. The combined extracorporeal blood purification method demonstrated similar efficacy in general ICU patients.

The aim of this study is to assess the efficiency and safety of combined extracorporeal blood purification in with septic shock in neurosurgical ICU in comparison with the efficiency and safety of the continuous renal replacement therapy (CRRT) with AN69 membrane.

Study novelty: We have not encountered published studies evaluating the efficiency of combined extracorporeal blood purification methods in neurosurgical patients with septic shock. Furthermore, currently there is not enough data to compare combined extracorporeal blood purification with CRRT for septic shock treatment. The planned study is the first to investigate the safety and efficiency of combined extracorporeal blood purification in patients with septic shock in neurosurgical ICU.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of septic shock according to SEPSIS 3 definition
* Glasgow Coma Scale of 4 and more on admission
* invasive hemodynamics monitoring
* norepinephrine > 0,1 µg/kg/min or use of 2 vasopressors

Exclusion Criteria:

* age <18 years
* >24 hours after diagnosis of septic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2021-09-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Vasopressor dose reduction | 6, 12, 24, 48 and 72 hours after the randomization time
  Vasopressor dose reduction value
Time on vasopressor support | Up to 28 days after the randomization date
  Time on vasopressor support
SOFA score reduction | 24, 48 and 72 hours after the randomization time
  SOFA score reduction

SECONDARY OUTCOMES:
Interleukins concentration reduction | 6, 12, 24 and 48 hours after the randomization time
  Interleukins (IL-1β, IL-6, IL-8, IL-10) concentration reduction
Tumor necrosis factor-α concentration reduction | 6, 12, 24 and 48 hours after the randomization time
  Tumor necrosis factor-α concentration reduction
Total bilirubin concentration reduction | 6, 12, 24 and 48 hours after the randomization time
  Total bilirubin concentration reduction
C - reactive protein level reduction | 24, 48 and 72 hours after the randomization time
  C - reactive protein level reduction
Procalcitonin concentration reduction | 6, 12, 24, 48 and 72 hours after the randomization time
  Procalcitonin concentration reduction
PiCCO-derived parameters normalization | 6, 12, 24, 48 and 72 hours after the randomization time
  Any PiCCO-derived parameter normalization
Arteriovenous pCO2 gap reduction | 6, 12, 24, 48 and 72 hours after the randomization time
  Arteriovenous pCO2 gap reduction
Arterial blood lactate level reduction | 6, 12, 24, 48 and 72 hours after the randomization time
  Arterial blood lactate level reduction
ICU length of stay | up to 3 months after the randomization date
  ICU length of stay
Hospital stay time | up to 3 months after the randomization date
  Hospital stay time
Mechanical ventilation time | up to 3 months after the randomization date
  Mechanical ventilation time
Continuous renal replacement therapy time | up to 3 months after the randomization date
  Continuous renal replacement therapy time

OTHER OUTCOMES:
Intracranial hemorrhagic complication | in 48 hours after the randomization time
  Presence of any intracranial hemorrhagic complications
Extracranial hemorrhagic complication | in 48 hours after the randomization time
  Presence of extracranial hemorrhagic complications
Death in 28-days after CRRT inititiation | 28-days after the randomization date
  28-days mortality in the observed sample group
In-hospital death | in 3 months after the randomization date
  Hospital mortality in the observed sample group
Albumin blood level reduction | 24 and 48 hours after the randomization time
  Albumin blood level reduction of more than 10%

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Burov, Study Chair — N. N. Burdenko National Medical Research Center of Neurosurgery
Locations (1):
- Federal State Autonomous Institution "N .N. Burdenko National Medical Research Center of Neurosurgery" of the Ministry of Healthcare of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No